CLINICAL TRIAL: NCT06860932
Title: A Palliative Care Model Impact on Knowledge and Attitudes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Aliza Bitton Ben-Zacharia, Assistant Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0535; UL1TR002384 (NIH)
Record Dates: First submitted 2025-02-05; First posted 2025-03-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis, MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Advance Directives

STUDY DESIGN:
Intervention Model Description: Guided by the Scott Murray's PC Transition Model, which integrates palliative services including decision making, communication, and coordinated care, the investigators will test the central hypothesis, and accomplish the objectives of this application by pursuing the following two specific aims in the pilot study:
  Aim 1: To explore the preferences of patients with neuroinflammatory diseases, PC knowledge, decisional conflict, and preparation for decision making among 50 adult (18-65 years) patients randomly assigned to one of two PC modalities: 1. a video depicting PC goals of care (intervention group, n=25), or 2. standard usual care using PC written information (control group, n=25).
  H1a: Patients randomized to the video will have higher documented preferences and fewer preferences for life-prolonging interventions (primary outcome) than the control group. The intervention group will have greater knowledge, lower decisional conflict, and greater preparation for decision making.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator): The control arm will follow standard of care which comprises palliative care (PC)written material about the PC conversation and advance directives.
  Interventions: Behavioral: Palliative care written material
- Intervention group (Active Comparator): The intervention group wil view a palliative care (PC) video discussing the PC conservation and advanced care planning (ACP).
  Interventions: Behavioral: Palliative care video comprises the conversation and advance directives.

INTERVENTIONS:
Behavioral: Palliative care video comprises the conversation and advance directives. — The palliative care video was done in a way that facilitates discussion and minimizes anxiety or any psychological risk/burden. The video is narrated by a young adult who opens with an empathic statement regarding the situation the young adult/adult patient finds themselves in. Then, there is a transition to contemplating what the future might hold and decisions about medical care and introducing the concept of ACP. There is acknowledgment that decision making is difficult, and that the presence of caregivers often helps. There is an explicit statement regarding values and spiritual beliefs and how that might impact decision making. The video then attempts to translate the preceding conversation into actionable medical orders using the most common three-goal framework that is based on the Physician Orders for Life Sustaining Treatment (POLST) paradigm: life-prolonging care, limited/blended care and comfort care.
  Arms: Intervention group
Behavioral: Palliative care written material — Written materials about palliative care conversation and advance directives.
  Arms: Control arm

SUMMARY:
This study is using a central, computer-generated simple randomization technique. Participants will be randomly assigned to groups within the constraints of ensuring balanced representation of gender, ethnicity, and race.

One-half of the patients are randomized to the decision aid video model, and one-half will serve as controls and receive a palliative care (PC) informational sheet. Sessions are designed to be consistent with PC principles of care using constructs from the Murray's transition theory including knowledge development coupled with advanced care planning (ACP)-to drive palliative care alongside curative treatment, and to support people with chronic progressive illnesses. The 2 groups will complete the demographic forms, and pre- and post-tests, at baseline and after three months. The intervention group will view the video decision aid, which takes 10 minutes, during their follow up appointment. The controls will read written information of the same content shown on the video and will complete similar questionnaires. The video opens with empathic statements regarding the situation in which patients may find themselves, including an introduction about medical decisions, and statements regarding values and spiritual beliefs and their impact on decision-making. The video translates the information into actionable medical orders using a three-goal framework: life-prolonging care, limited/blended care, and comfort care. The video describes the features of each of the goals of care and the risks and benefits of each option using visual images that illustrate the interventions. Patients will review the video using iPads and will be able to review the video again as needed. The Flesch-Kincaid ease score for the video narration is 71.6; for the "Conversation" piece, it is 65.9. These indicate that the passages require approximately a 7th or 8th grade reading level, which Flesch suggests makes them "easy to read" and "plain English," respectively.

The goal of the video intervention is to help patients express their values and health goals, while achieving their life and core values. The intervention group will view the video which includes modules to teach patients strategies for expressing their concerns and enhance their self-efficacy, helping them overcome any barriers. To enhance intervention fidelity, an ACP facilitator guide will be developed as reference for the intervention implementation. It will detail the key topics and purposes of each session of the intervention, the guiding questions, and the facilitation skills.

Aim 1: To explore the preferences of patients with neuroinflammatory diseases, PC knowledge, decisional conflict, and preparation for decision making among 50 adult (18-65 years old) patients randomly assigned to one of two PC modalities: 1. a video depicting PC goals of care (intervention group, n=25), or 2. standard usual care using PC written information (control group, n=25).

H1a: Patients randomized to the video will have higher documented preferences and fewer preferences for life-prolonging interventions (primary outcome) than the control group. The intervention group will have greater knowledge, lower decisional conflict, and greater preparation for decision making than those randomized to the control group.

Aim 2: To compare PC conversations and documentation at 3 months among patients with neuroinflammatory diseases.

H2: Patients randomized to the video will have more PC conversations and higher rates of PC documentation after 3 months.

DETAILED DESCRIPTION:
Patients will be asked for their goals-of-care preferences at baseline, after watching the video or reading the information sheet and after three months. Patients will be asked for their goals-of-care preference (Life-prolonging, Limited/Blended, Comfort, or Unsure), cardiopulmonary resuscitation (CPR) preference (Yes, No, or Unsure), and ventilatory support (Yes, No, or Unsure) at baseline, and then again immediately after watching the video or reviewing the informational sheet, and then the investigators will contact all patients after 3 months by telephone to ask for their preferences again. The investigators will also have an open-ended question for those subjects who change their preferences from the initial post-video or control survey ("Can patients tell us more about why they have changed their preference from the one stated before?"). The primary outcome is patient treatment preferences (i.e., care considerations, discontinuation of care, versus continued full care) for neurological care (Aim 1). The preferences will be measured as a binary outcome based on our clinical experience. When a patient chooses "" as an option for any of the treatment outcomes, in clinical care that is equivalent to the default (i.e., full code or life-prolonging interventions). Secondary outcomes include knowledge, decisional conflict, and preparation for decision making (Aims 1). The investigators will also explore the stability of preferences and documentation after 3 months (Aim 2). In all of investigators' prior trials, 3 months has been the requisite amount of time needed for patients to contemplate their decisions regarding medical care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MS, NMOSD, or anti-MOG, at least 2 years after their diagnosis.
* Aged 18-65
* Speak English since all instruments are available in English.

Exclusion Criteria:

* Visually impaired (note, hearing impaired is not an exclusion criterion as the video is closed captioned).
* Psychological state not appropriate for PC discussions as determined by the Patient Health Questionnaire 9 (PHQ9).
* A score of 11 or higher, indicative of major depressive disorder, will be referred to immediate management and excluded from the study.
* Unable to participate in PC discussions due to cognitive impairment as determined by the Processing Speed Test (PST) score below -1.5 Z score.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Palliative care preferences (i.e., care considerations, discontinuation of care, versus continued full care) for neurological care (Aim 1). | 3 months.
  The patient treatment preferences (i.e., care considerations, discontinuation of care, versus continued full care) for neurological care. The preferences will be measured based on a questionnaire asking patients about their preferences after viewing the PC video or reading the written material.

SECONDARY OUTCOMES:
Palliative care knowledge | 3 months
  The palliative care knoeldge will be assessed using the palliative care knowledge scale (PaCKS). This scale has 13 questions on palliative care definitions and goals.
Preparation for decision making | 3 months
  The investigators will assess patients/care partners' perception of how useful a decision aid is in communicating and making decisions using the well-validated Preparation for Decision Making Scale.
Decisional conflict | 3 months.
  The Decision Conflict validated scale measures uncertainty regarding decision making associated with palliative care.
Advance care planning engagement | 3 months.
  Advance care planning (ACP) engagement: The investigators will use the ACPE 15 questions tool about engagement, which is a well-validated tool.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Judith Jaffe Multiple Sclerosis Center, New York, New York
  - Hunter College, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ben-Zacharia AB, Bethoux FA, Volandes A. Self-Perceived Knowledge and Comfort Discussing Palliative Care and End-of-Life Issues among Professionals Managing Neuroinflammatory Diseases. J Palliat Med. 2021 May;24(5):725-735. doi: 10.1089/jpm.2020.0268. Epub 2020 Oct 16. PMID 33064605
- [Background] Ben-Zacharia AB, Brugger HT, Carbone S, Malchiodi J, Wallace E, Bethoux F, Volandes A, Bartels A. Palliative Care Knowledge and Attitudes Among Patients With Neuroinflammatory Diseases. J Palliat Med. 2024 Jan;27(1):10-17. doi: 10.1089/jpm.2023.0224. Epub 2023 Aug 22. PMID 37610856